CLINICAL TRIAL: NCT05959629
Title: A Clinical Use of Er,Cr:YSGG Laser: an Anti-biofilm Treatment
Brief Title: Erbium, Chromium: Yttrium, Scandium, Gallium, Garnet (Er,Cr:YSGG) Laser in Root Canal Disinfection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to follow up participants due to geographic location and other reasons.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 853701
Record Dates: First submitted 2023-07-05; First posted 2023-07-25 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Endodontic Disease; Root Canal Infection
Keywords: Root Canal Irrigants; lasers
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Sodium Hypochlorite

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Waterlase Express™, BIOLASE® (Experimental): Root canals will be instrumented up to size 30/0.04 taper using Er,Cr:YSGG laser (Waterlase Express™, BIOLASE®), followed by standard of care (NaOCl).
  Interventions: Device: Waterlase Express™, BIOLASE®
- Sodium Hypochlorite (Active Comparator): Root canals will be instrumented up to size 30/0.04 taper using standard of care (NaOCl).
  Interventions: Other: Sodium Hypochlorite

INTERVENTIONS:
Device: Waterlase Express™, BIOLASE® — Er,Cr:YSGG laser 2780nm (Waterlase Express™, BIOLASE®) with 300μm tip (EdgePro #3) will be placed into the mid-root of the canal. The tip will be activated and slowly withdrawn to the orifice (1-2mm/sec) following the manufacturer settings (energy 15 Millijoule (mJ), repetition rate 50 Hertz (Hz), 0% air, 0% water).
  Other Names: Er,Cr:YSGG laser; Waterlase Express™
  Arms: Waterlase Express™, BIOLASE®
Other: Sodium Hypochlorite — Root canals will be instrumented up to size 30/0.04 taper using 1.5cc of 3% NaOCl in between files.
  Other Names: NaOCl
  Arms: Sodium Hypochlorite

SUMMARY:
The purpose of this study is to develop a protocol for biofilms disinfection with a FDA cleared, clinically approved and commercially available Er,Cr:YSGG laser treatments. This protocol will be testing local single topical application of Lasers within the canal system in patients going through routine endodontic treatment, evaluate its potential as anti-biofilm treatment and compare it to other currently used antibacterial protocols.

DETAILED DESCRIPTION:
After being informed about the study and its potential risk, for all patients giving written informed consent we will screen potential participants by inclusion and exclusion criteria; clinical assessment, obtain radiographs, medical history/medications and documents to determine eligibility for study entry. Participants who meet the eligibility requirements will be randomized in a 1:1 ratio to Group 1: Standard of care irrigation protocol "Sodium Hypochlorite (NaOCl)", Group 2: Er,Cr:YSGG laser + standard of care irrigation protocol (NaOCl).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female (Gender is not an inclusion or exclusion criteria), aged 18 years old or above.
* In good general health as evidenced by medical history or non-contributory medical history (Patient can be seen for regular dental appointment in Penn Dental Medicine; American Society of Anesthesiologists (ASA) classes I and II).
* Radiographic presence of periapical radiolucency.
* Negative response to thermal sensitivity testing (difluorochloromethane at -50 °C, Endo-Ice, Coltène/Whaledent Inc., Cuyahoga Falls, Ohio) or electric pulp testing.
* Enough tooth structure for adequate isolation with rubber dam.
* No history of previous endodontic treatment on the tooth.
* Teeth with single canal, 1 distal canal of lower molar, 1 palatal canal of upper molar.

Exclusion Criteria:

* Patients who report they are pregnant.
* Teeth affected by dental trauma.
* Periodontal changes (pockets 3 mm, mobility I or gingival edema).
* Radiographic presence of resorptive processes.
* Per the investigator's discretion, unable or unlikely to comply with study procedure.
* Presence of any condition which, in the opinion of the investigator, makes participation in the study not in the individual's best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bekir Karabucak, DMD, MS., Principal Investigator — Chair and Professor of Endodontics. Postdoctoral Endodontics Program, Director.; Flavia Teles, DDS,MS,DMSc, Principal Investigator — Associate Professor, Department of Basic & Translational Sciences
Locations (1):
- University of Pennsylvania, School of Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu YH, Kushnir L, Kohli M, Karabucak B. Comparing the incidence of postoperative pain after root canal filling with warm vertical obturation with resin-based sealer and sealer-based obturation with calcium silicate-based sealer: a prospective clinical trial. Clin Oral Investig. 2021 Aug;25(8):5033-5042. doi: 10.1007/s00784-021-03814-x. Epub 2021 Feb 8. PMID 33555456
- [Background] Orstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Endod Dent Traumatol. 1986 Feb;2(1):20-34. doi: 10.1111/j.1600-9657.1986.tb00119.x. No abstract available. PMID 3457698
- [Background] KAKEHASHI S, STANLEY HR, FITZGERALD RJ. THE EFFECTS OF SURGICAL EXPOSURES OF DENTAL PULPS IN GERM-FREE AND CONVENTIONAL LABORATORY RATS. Oral Surg Oral Med Oral Pathol. 1965 Sep;20:340-9. doi: 10.1016/0030-4220(65)90166-0. No abstract available. PMID 14342926
- [Background] Bergenholtz G. Micro-organisms from necrotic pulp of traumatized teeth. Odontol Revy. 1974;25(4):347-58. No abstract available. PMID 4155793
- [Background] Kerekes K, Tronstad L. Long-term results of endodontic treatment performed with a standardized technique. J Endod. 1979 Mar;5(3):83-90. doi: 10.1016/S0099-2399(79)80154-5. No abstract available. PMID 296248
- [Background] Sjogren U, Figdor D, Persson S, Sundqvist G. Influence of infection at the time of root filling on the outcome of endodontic treatment of teeth with apical periodontitis. Int Endod J. 1997 Sep;30(5):297-306. doi: 10.1046/j.1365-2591.1997.00092.x. PMID 9477818
- [Background] Bystrom A, Sundqvist G. The antibacterial action of sodium hypochlorite and EDTA in 60 cases of endodontic therapy. Int Endod J. 1985 Jan;18(1):35-40. doi: 10.1111/j.1365-2591.1985.tb00416.x. No abstract available. PMID 3922900
- [Background] Bystrom A, Sundqvist G. Bacteriologic evaluation of the effect of 0.5 percent sodium hypochlorite in endodontic therapy. Oral Surg Oral Med Oral Pathol. 1983 Mar;55(3):307-12. doi: 10.1016/0030-4220(83)90333-x. PMID 6572884
- [Background] Bystrom A, Sundqvist G. Bacteriologic evaluation of the efficacy of mechanical root canal instrumentation in endodontic therapy. Scand J Dent Res. 1981 Aug;89(4):321-8. doi: 10.1111/j.1600-0722.1981.tb01689.x. PMID 6947391
- [Background] Nair PN, Henry S, Cano V, Vera J. Microbial status of apical root canal system of human mandibular first molars with primary apical periodontitis after "one-visit" endodontic treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Feb;99(2):231-52. doi: 10.1016/j.tripleo.2004.10.005. PMID 15660098
- [Background] Ricucci D, Siqueira JF Jr, Bate AL, Pitt Ford TR. Histologic investigation of root canal-treated teeth with apical periodontitis: a retrospective study from twenty-four patients. J Endod. 2009 Apr;35(4):493-502. doi: 10.1016/j.joen.2008.12.014. PMID 19345793
- [Background] Vera J, Siqueira JF Jr, Ricucci D, Loghin S, Fernandez N, Flores B, Cruz AG. One- versus two-visit endodontic treatment of teeth with apical periodontitis: a histobacteriologic study. J Endod. 2012 Aug;38(8):1040-52. doi: 10.1016/j.joen.2012.04.010. Epub 2012 Jun 12. PMID 22794203
- [Background] Ricucci D, Siqueira JF Jr. Biofilms and apical periodontitis: study of prevalence and association with clinical and histopathologic findings. J Endod. 2010 Aug;36(8):1277-88. doi: 10.1016/j.joen.2010.04.007. Epub 2010 Jun 14. PMID 20647081
- [Background] Zorita-Garcia M, Alonso-Ezpeleta LO, Cobo M, Del Campo R, Rico-Romano C, Mena-Alvarez J, Zubizarreta-Macho A. Photodynamic therapy in endodontic root canal treatment significantly increases bacterial clearance, preventing apical periodontitis. Quintessence Int. 2019;50(10):782-789. doi: 10.3290/j.qi.a43249. PMID 31559398
- [Background] Wang X, Cheng X, Liu B, Liu X, Yu Q, He W. Effect of Laser-Activated Irrigations on Smear Layer Removal from the Root Canal Wall. Photomed Laser Surg. 2017 Dec;35(12):688-694. doi: 10.1089/pho.2017.4266. Epub 2017 Apr 5. PMID 28394240
- [Background] Bordea IR, Hanna R, Chiniforush N, Gradinaru E, Campian RS, Sirbu A, Amaroli A, Benedicenti S. Evaluation of the outcome of various laser therapy applications in root canal disinfection: A systematic review. Photodiagnosis Photodyn Ther. 2020 Mar;29:101611. doi: 10.1016/j.pdpdt.2019.101611. Epub 2019 Dec 3. PMID 31809911
- [Background] Meire MA, Coenye T, Nelis HJ, De Moor RJ. Evaluation of Nd:YAG and Er:YAG irradiation, antibacterial photodynamic therapy and sodium hypochlorite treatment on Enterococcus faecalis biofilms. Int Endod J. 2012 May;45(5):482-91. doi: 10.1111/j.1365-2591.2011.02000.x. Epub 2012 Jan 14. PMID 22243483
- [Background] Josic U, Mazzitelli C, Maravic T, Fidler A, Breschi L, Mazzoni A. Biofilm in Endodontics: In Vitro Cultivation Possibilities, Sonic-, Ultrasonic- and Laser-Assisted Removal Techniques and Evaluation of the Cleaning Efficacy. Polymers (Basel). 2022 Mar 25;14(7):1334. doi: 10.3390/polym14071334. PMID 35406207
- [Background] Seet AN, Zilm PS, Gully NJ, Cathro PR. Qualitative comparison of sonic or laser energisation of 4% sodium hypochlorite on an Enterococcus faecalis biofilm grown in vitro. Aust Endod J. 2012 Dec;38(3):100-6. doi: 10.1111/j.1747-4477.2012.00366.x. Epub 2012 Jul 16. PMID 23211068
- [Background] Suer K, Ozkan L, Guvenir M. Antimicrobial effects of sodium hypochlorite and Er,Cr:YSGG laser against Enterococcus faecalis biofilm. Niger J Clin Pract. 2020 Sep;23(9):1188-1193. doi: 10.4103/njcp.njcp_632_18. PMID 32913155
- [Background] Martins MR, Carvalho MF, Pina-Vaz I, Capelas JA, Martins MA, Gutknecht N. Outcome of Er,Cr:YSGG laser-assisted treatment of teeth with apical periodontitis: a blind randomized clinical trial. Photomed Laser Surg. 2014 Jan;32(1):3-9. doi: 10.1089/pho.2013.3573. Epub 2013 Dec 13. PMID 24328607
- [Background] Dalton BC, Orstavik D, Phillips C, Pettiette M, Trope M. Bacterial reduction with nickel-titanium rotary instrumentation. J Endod. 1998 Nov;24(11):763-7. doi: 10.1016/S0099-2399(98)80170-2. PMID 9855830
- [Background] Shuping GB, Orstavik D, Sigurdsson A, Trope M. Reduction of intracanal bacteria using nickel-titanium rotary instrumentation and various medications. J Endod. 2000 Dec;26(12):751-5. doi: 10.1097/00004770-200012000-00022. PMID 11471648
- [Background] McGurkin-Smith R, Trope M, Caplan D, Sigurdsson A. Reduction of intracanal bacteria using GT rotary instrumentation, 5.25% NaOCl, EDTA, and Ca(OH)2. J Endod. 2005 May;31(5):359-63. doi: 10.1097/01.don.0000145035.85272.7c. PMID 15851929
- [Background] Wang CS, Arnold RR, Trope M, Teixeira FB. Clinical efficiency of 2% chlorhexidine gel in reducing intracanal bacteria. J Endod. 2007 Nov;33(11):1283-9. doi: 10.1016/j.joen.2007.07.010. PMID 17963947

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Allocated to control: n=28, received allocated control =26. 2 when accessed were partially necrotic.
  Allocated to intervention: n=28, received allocated control =26. 2 had technical issues.
Period: Overall Study
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Started | 28 | 28
Completed | 26 | 26
Not Completed | 2 | 2
Not completed — partially necrotic/technical issues | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 52
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (2) | 44.125 (2) | 44.57 (2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: participants included in the study
  Participants
    Female | 13 | 13 | 26
    Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 26 | 26 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: The Change in Bacterial Count Between the Experimental Group (Laser) and the Standard of Care (NaOCl) Group (Routinely Used Irrigation Protocol).
Description: By measuring change in bacteria colony forming units (CFU) before and after treatment for the experimental group (laser) and the standard of care (NaOCl) group, then comparing the two groups.
Time Frame: All samples will be taken during the first root canal treatment visit. Sample1 before cleaning or shaping the root canal.
Measure: Mean (Standard Deviation); unit: Mean CFU
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 26 | 26
Mean CFU | 8.279923256 (2.933726699) | 8.601200494 (2.99841829)

2. Primary Outcome: The Change in Bacterial Count Between the Experimental Group (Laser) and the Standard of Care (NaOCl) Group (Routinely Used Irrigation Protocol).
Description: as for outcome 1
Time Frame: All samples will be taken during the first root canal treatment visit. Sample2 after cleaning and shaping of the root canal using laser or NaOCl.
Measure: Mean (Standard Deviation); unit: Mean CFU
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 26 | 26
Mean CFU | 4.332058015 (2.154027598) | 4.373858908 (2.532760244)

3. Primary Outcome: The Change in Bacterial Count Between the Experimental Group (Laser) and the Standard of Care (NaOCl) Group (Routinely Used Irrigation Protocol).
Description: By measuring change in bacteria colony forming units (CFU) before and after treatment for the experimental group (laser) and the standard of care (NaOCl) group, then completion of final routine irrigation protocol, then comparing the two groups.
Time Frame: All samples will be taken during the first root canal treatment visit. Sample 3 Upon completion of final routine irrigation protocol.
Measure: Mean (Standard Deviation); unit: Mean CFU
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 26 | 26
Mean CFU | 2.765533576 (2.087467581) | 2.570435011 (2.413322255)

4. Secondary Outcome: Mean Change From Baseline in Pain Scores at 4-hours After the Procedure on a Numeric Rating Scale (NRS)
Description: Following a previous published study done at the Department of Endodontics, University of Pennsylvania. Patients will be asked to rate the intensity of preoperative pain on a numeric rating scale (NRS) from 0 (no pain) to 10 (worst pain) before receiving root canal treatment. Along with NRS, the Wong-Baker facial grimace scale (images) will also be presented to the patients to help them in scoring the pain.
  Patients will be asked to rate the intensity of postoperative pain at 4-hours after the procedure.
  Change = (4 hours score - baseline score)
Time Frame: At the end of the first root canal treatment visit, patients will be given a survey and asked to rate the intensity of preoperative pain and postoperative pain at 4-hours post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 26 | 26
units on a scale
  t0 | 3.28 (3.67) | 2.38 (3.68)
  t4 | 3.32 (2.67) | 2.67 (2.66)

5. Secondary Outcome: Secondary Outcome: Mean Change From Baseline in Pain Scores at 24 Hours After the Procedure on a Numeric Rating Scale (NRS).
Description: Following a previous published study done at the Department of Endodontics, University of Pennsylvania. Patients will be asked to rate the intensity of preoperative pain on a numeric rating scale (NRS) from 0 (no pain) to 10 (worst pain) before receiving root canal treatment. Along with NRS, the Wong-Baker facial grimace scale (images) will also be presented to the patients to help them in scoring the pain.
  Patients will be asked to rate the intensity of postoperative pain at 24-hours after the procedure.
  Change = (24 hours score - baseline score)
Time Frame: At the end of the first root canal treatment visit, patients will be given a survey and asked to rate the postoperative pain at 24-hours post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 26 | 26
score on a scale | 2.16 (2.62) | 1.13 (1.92)

6. Secondary Outcome: Mean Change From Baseline in Pain Scores at 48-hours After the Procedure on a Numeric Rating Scale (NRS)
Description: Following a previous published study done at the Department of Endodontics, University of Pennsylvania. Patients will be asked to rate the intensity of preoperative pain on a numeric rating scale (NRS) from 0 (no pain) to 10 (worst pain) before receiving root canal treatment. Along with NRS, the Wong-Baker facial grimace scale (images) will also be presented to the patients to help them in scoring the pain.
  Patients will be asked to rate the intensity of postoperative pain at 48-hours after the procedure.
  Change = (48 hours score - baseline score)
Time Frame: At the end of the first root canal treatment visit, patients will be given a survey and asked to rate the postoperative pain at 48-hours post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 26 | 26
score on a scale | 1.44 (0.58) | 2.20 (1.50)

7. Secondary Outcome: Periapical Bone Changes From Baseline in Periapical Radiographs at 6 Months Follow Up
Description: Periapical radiographs will be taken at baseline (preoperative) then at 6 months follow up post root canal filling
  Radiographically, Following periapical index (PAI) by Órstavik 1986, description of radiographic findings:
  1. Normal periapical structures.
  2. Small changes in the bone structure.
  3. Change in the bone structure with mineral loss.
  4. Periodontitis with a well-defined radiolucent area.
  5. Severe periodontitis with exacerbating features.
  Success is defined as either complete (radiographic resolution of a periapical lesion - the radiographic sign of inflammatory processes surrounding a root tip) or incomplete healing (scar tissue formation) and failure includes uncertain healing (radiographic reduction of a periapical lesion or same lesion size) or unsatisfactory healing (increase in lesion size) as determined on the radiograph.
Time Frame: Periapical bone changes measured at baseline and 6 months follow up (± 7 days) post root canal filling.
Population: The study was terminated. Data were not collected for this measure at any time point.
  Unable to follow up participants due to their geographic location and other reasons.
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Periapical Bone Changes From Baseline in Periapical Radiographs at 1 Year Follow Up
Description: Periapical radiographs will be taken at baseline (preoperative) then at 1 year follow up post root canal filling
  Radiographically, Following periapical index (PAI) by Órstavik 1986, description of radiographic findings:
  1. Normal periapical structures.
  2. Small changes in the bone structure.
  3. Change in the bone structure with mineral loss.
  4. Periodontitis with a well-defined radiolucent area.
  5. Severe periodontitis with exacerbating features.
  Success is defined as either complete (radiographic resolution of a periapical lesion - the radiographic sign of inflammatory processes surrounding a root tip) or incomplete healing (scar tissue formation) and failure includes uncertain healing (radiographic reduction of a periapical lesion or same lesion size) or unsatisfactory healing (increase in lesion size) as determined on the radiograph.
Time Frame: Periapical bone changes measured at baseline and 1 year follow up (± 7 days) post root canal filling.
Population: as for outcome 7
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Periapical Bone Changes From Baseline in Periapical Radiographs at 2 Years Follow Up
Description: Periapical radiographs will be taken at baseline (preoperative) then at 2 years follow up post root canal filling
  Radiographically, Following periapical index (PAI) by Órstavik 1986, description of radiographic findings:
  1. Normal periapical structures.
  2. Small changes in the bone structure.
  3. Change in the bone structure with mineral loss.
  4. Periodontitis with a well-defined radiolucent area.
  5. Severe periodontitis with exacerbating features.
  Success is defined as either complete (radiographic resolution of a periapical lesion - the radiographic sign of inflammatory processes surrounding a root tip) or incomplete healing (scar tissue formation) and failure includes uncertain healing (radiographic reduction of a periapical lesion or same lesion size) or unsatisfactory healing (increase in lesion size) as determined on the radiograph.
Time Frame: Periapical bone changes measured at baseline and 2 years follow up (± 7 days) post root canal filling.
Population: as for outcome 7
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Presence of Clinical Signs or Symptoms at 6 Months Follow Up
Description: Clinical signs and symptoms: Pain, swelling, percussion sensitivity and sinus tracts measured at 6 months follow up.
  Clinically success is defined by the absence of pain, swelling, percussion sensitivity or sinus tracts.
  Clinical failure is defined as the persistent presence of any of the signs and symptoms mentioned above.
Time Frame: Clinical signs and symptoms measured at 6 months (± 7 days) post root canal filling.
Population: as for outcome 7
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Presence of Clinical Signs or Symptoms at 1 Year Follow Up
Description: Clinical signs and symptoms: Pain, swelling, percussion sensitivity and sinus tracts measured at 1 year follow up.
  Clinically success is defined by the absence of pain, swelling, percussion sensitivity or sinus tracts.
  Clinical failure is defined as the persistent presence of any of the signs and symptoms mentioned above.
Time Frame: Clinical signs and symptoms measured at 1 year (± 7 days) post root canal filling.
Population: as for outcome 7
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Presence of Clinical Signs or Symptoms at 2 Years Follow Up
Description: Clinical signs and symptoms: Pain, swelling, percussion sensitivity and sinus tracts measured at 2 years follow up.
  Clinically success is defined by the absence of pain, swelling, percussion sensitivity or sinus tracts.
  Clinical failure is defined as the persistent presence of any of the signs and symptoms mentioned above.
Time Frame: Clinical signs and symptoms measured at 2 years (± 7 days) post root canal filling.
Population: as for outcome 7
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Tooth Survival at 6 Months Follow Up
Description: Tooth survival is defined as the presence of the tooth inside the mouth.
  Success: Tooth is still present in the oral cavity. Failure: Tooth is extracted for any reason.
Time Frame: Measured at 6 months (± 7 days) post root canal filling.
Population: as for outcome 7
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Tooth Survival at 1 Year Follow Up
Description: as for outcome 13
Time Frame: Measured at 1 year (± 7 days) post root canal filling.
Population: as for outcome 7
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Tooth Survival at 2 Years Follow Up
Description: as for outcome 13
Time Frame: Measured at 2 years (± 7 days) post root canal filling.
Population: as for outcome 7
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Waterlase Express™, BIOLASE® | Sodium Hypochlorite
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT05959629/Prot_SAP_000.pdf